CLINICAL TRIAL: NCT01419561
Title: Natural History Study of the KSHV Inflammatory Cytokine Syndrome (KICS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110220; 11-C-0220
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-11

CONDITIONS: KSHV Inflammatory Cytokine Syndrome (KICS); KSHV; HHV-8
Keywords: KSHV; KICS; HIV; Cytokines; HHV-8
MeSH Terms: interventions — Zidovudine; liposomal doxorubicin; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1 (No Intervention): Evaluation for Alternative Causes of KICS Symptoms (inactive)
- 2 (No Intervention): Natural history/Observation arm (inactive)
- 3 (Experimental): High dose zidovudine + valganciclovir (inactive)
  Interventions: Drug: Zidovudine; Drug: Valganiclovir
- 4 (Experimental): Rituximab with or without liposomal doxorubicin (inactive)
  Interventions: Drug: Liposomal Doxorubicin; Drug: Rituximab
- 5 (Other): Standard and alternative rational therapies (inactive)
  Interventions: Other: Standard Therapies
- 6 (Other): Natural history
  Interventions: Other: Cohort 1

INTERVENTIONS:
Drug: Zidovudine — Zidovudine 600 mg will be administered orally 4 times a day or i.v. at 300 mg every 6 hours for 14 days for cycle 1 and for 7 days (up to additional 7 days if ongoing symptoms) for following cycles.
  Arms: 3
Drug: Liposomal Doxorubicin — Liposomal doxorubicin (20 mg/m2) will be administered i.v. over 1 hour at day 1 of each cycle
  Arms: 4
Drug: Valganiclovir — Valganciclovir (900mg) will be administered orally twice/day or Ganciclovir (5 mg/kg) will be administered i.v. over 1 hour for 14 days for cycle 1 and for 7 days (up to additional 7 days if ongoing symptoms) for following cycles.
  Arms: 3
Drug: Rituximab — Rituximab (375 mg/m2) will be admnistered i.v. at 50 mg/hr up to 100 mg/hr at day 1 of the first cycle and at 100mg/hr up to 400 mg
  /hr at day 1 of following cycles.
  Arms: 4
Other: Standard Therapies — Standard of Care drugs
  Arms: 5
Other: Cohort 1 — Participants who are infected with KSHV who meet criteria for inflammatory cytokine syndrome (KICS)
  Arms: 6

SUMMARY:
Background:

- KSHV inflammatory cytokine syndrome (KICS) is a newly recognized disease caused by Kaposi sarcoma-associated herpesvirus (KSHV). This virus can cause cancer. People with KICS can have severe symptoms. They include fever, weight loss, and fluid in the legs or abdomen. People with KICS may also be at risk of getting other cancers associated with KSHV. These cancers include Kaposi sarcoma and lymphoma. Because KICS is a newly identified disease, more information is needed on how the disease works and what can be done to treat it.

Objectives:

- To collect genetic and medical information from people with KSHV inflammatory cytokine syndrome.

Eligibility:

- Individuals at least 18 years of age who have Kaposi sarcoma herpes virus and symptoms that resemble those caused by KICS.

Design:

* Participants will have regular study visits. The schedule will be determined by the study researchers.
* Participants will provide a complete medical history and have a full physical exam. Blood and urine samples will be collected as well.
* People with KICS that requires treatment may get new experimental treatments. These treatments may include antiviral drugs and chemotherapy drugs, depending on the nature of the disease.
* Participants will have imaging studies, such as chest x-rays and computed tomography scans, to study the tumors.
* Bone marrow and lymph node biopsies may be done to collect tissue samples for study.
* Participants who have Kaposi sarcoma will have photographs taken of their lesions....

DETAILED DESCRIPTION:
Background

-Kaposi sarcoma-associated herpesvirus (KSHV) inflammatory cytokine syndrome (KICS) is a newly recognized syndrome caused by KSHV. It is characterized by severe inflammatory symptoms including fevers, wasting, cytopenias, hypoalbuminemia, and hyponatremia, associated in some cases with lymphadenopathy or effusions, without pathological evidence of MCD. Patients with KICS exhibit elevated KSHV viral loads and cytokine dysregulation, with elevations of IL-6, IL-10, and a KSHV-encoded IL-6 homolog, viral IL-6.

Objective

-Assessment of the natural history of KSHV inflammatory cytokine syndrome (KICS), including the spectrum of clinical, laboratory and radiographic abnormalities seen in affected participants.

Eligibility

* Adults of any HIV status with:

  * At least two symptoms, laboratory or radiographic abnormalities which are at least possibly attributable to KICS (including fever, fatigue, cachexia, edema, respiratory or gastrointestinal symptoms, hematologic cytopenias, hypoalbuminemia, hyponatremia, lymphadenopathy, organomegaly, effusions)
  * C-reactive protein >3mg/L
  * Evidence of KSHV infection or a risk exposure for KSHV infection
  * No evidence of KSHV-associated multicentric Castleman disease
* Participants with these characteristics will be further evaluated to identify those whose clinical and laboratory features are consistent with the KICS working case definition to be followed in the natural history phase of the study.

Design

-This is a single center natural history study with a cohort of up to 120 evaluable participants. Participants who meet the criteria for KICS will go onto a natural history arm, which permits observation for KICS with or without other concurrent KSHV-associated disorders. Participants who require KS and/or primary effusion lymphoma (PEL) treatment along with a KICS diagnosis will receive rational therapies for these conditions or be treated for their KS and/or PEL on a separate protocol while still followed on this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to18 Years.
* Any HIV status.
* At least two manifestations drawn from at least two of the categories (clinical symptoms, laboratory abnormalities and/or radiographic abnormalities), which are at least possibly attributable to KICS and are not readily explicable from known medical conditions in the participant:
* Clinical symptoms (each at least grade 1 by CTCAE definitions)
* Fever (>38 degrees C), chills or rigors
* Fatigue or lethargy
* Cachexia or edema
* Cough, dyspnea, airway hyperreactivity, or nasal inflammation
* Nausea, anorexia, abdominal pain or altered bowel habit
* Athralgia or myalgia
* Altered mental state
* Neuropathy with or without pain
* Laboratory abnormalities
* Anemia (hemoglobin<12.0g/dL)
* Thrombocytopenia (platelets<100,000 cells/microL)
* Leukopenia (white cell count<4,000 cells/microL)
* Hypoalbuminemia (albumin<3.5g/dL)
* Hyponatremia (sodium<135mmol/L)
* Coagulopathy (PT or PTT >1.5 times upper limit of normal)
* Radiographic Abnormalities
* Pathologic lymphadenopathy (at least five discrete nodes each >1cm in their longest dimension)
* Splenomegaly (>12 cm in the longest dimension)
* Hepatomegaly (>17cm in the longest dimension)
* Body cavity effusions not caused by primary effusion lymphoma nor chylous effusions directly related to lymphatic infiltration by KS
* C-reactive protein (CRP) >3mg/L.
* Exposure risk for KSHV infection (including being a first or second generation immigrant from an endemic area, or male-to-male sexual activity) or evidence of KSHV infection demonstrated by one of:

  * Molecular evidence of KSHV in whole blood, or KSHV VL levels within circulating PBMCs as determined by the Whitby laboratory
  * Immunohistochemical evidence of KSHV in tissues (for example by staining for LANA or vIL-6) confirmed in the Laboratory of Pathology (LP), CCR, NCI.
  * Presence of KS or PEL (KSHV-associated malignancies), confirmed in the LP, CCR, NCI.
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and after treatment (if received), according to drug requirements. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

- Biopsy proven KSHV-associated MCD, confirmed in the LP, CCR, NCI.

Note: In collaboration with LP, we have recently found that some participants with KICS but without a lymph node or splenic diagnosis of MCD have MCD-like cells in their effusions or circulating blood. This may in fact represent a newly recognized form of KSHV-MCD, but our analysis continues. While certain of these participants were historically included in this study, given this new understanding, they will not be entered on this protocol and removed if liquid MCD is diagnosed.

* Pregnancy
* Any abnormality that would be scored as NCI CTC Grade 4 toxicity that is unrelated to HIV, its treatment, or to KICS that would preclude the use of all of the study treatments or the ability to monitor the natural history of KICS untreated.
* Any condition or set of circumstances that in the opinion of the investigators would make participation in this study unsafe or otherwise inappropriate for a given individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-09-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Natural history of KICS | one year
  Description of the natural history of KICS, including the spectrum of clinical, laboratory and radiographic abnormalities seen in affected patients

SECONDARY OUTCOMES:
Participants with KICS | one year
  Evaluate the survival of participants with KICS and of KICS with primary effusion lymphoma (PEL)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chang Y, Cesarman E, Pessin MS, Lee F, Culpepper J, Knowles DM, Moore PS. Identification of herpesvirus-like DNA sequences in AIDS-associated Kaposi's sarcoma. Science. 1994 Dec 16;266(5192):1865-9. doi: 10.1126/science.7997879.
- [Background] Moore PS, Gao SJ, Dominguez G, Cesarman E, Lungu O, Knowles DM, Garber R, Pellett PE, McGeoch DJ, Chang Y. Primary characterization of a herpesvirus agent associated with Kaposi's sarcomae. J Virol. 1996 Jan;70(1):549-58. doi: 10.1128/JVI.70.1.549-558.1996. PMID 8523568
- [Background] Viejo-Borbolla A, Schulz TF. Kaposi's sarcoma-associated herpesvirus (KSHV/HHV8): key aspects of epidemiology and pathogenesis. AIDS Rev. 2003 Oct-Dec;5(4):222-9. PMID 15012001
- [Derived] Ramaswami R, Lurain K, Polizzotto MN, Widell A, Ekwede I, Tassi E, Rupert A, Marshall VA, Roth MJ, Filie AC, Pittaluga S, Jaffe ES, Wang HW, Whitby D, Uldrick TS, Yarchoan R. Characteristics and outcomes of Kaposi sarcoma herpesvirus-associated inflammatory cytokine syndrome. Blood Adv. 2025 Nov 25;9(22):5720-5731. doi: 10.1182/bloodadvances.2025016685. PMID 40763275
- [Derived] Lage SL, Ramaswami R, Rocco JM, Rupert A, Davis DA, Lurain K, Manion M, Whitby D, Yarchoan R, Sereti I. Inflammasome activation in patients with Kaposi sarcoma herpesvirus-associated diseases. Blood. 2024 Oct 3;144(14):1496-1507. doi: 10.1182/blood.2024024144. PMID 38941593
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-C-0220.html